CLINICAL TRIAL: NCT00005350
Title: Evaluating Strategies to Control Hypercholesterolemia
Status: Completed | Type: Observational
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4219; R01HL046297 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia

SUMMARY:
To determine the cost-effectiveness of alternative strategies for cholesterol reduction.

DETAILED DESCRIPTION:
BACKGROUND:

The availability of effective treatment for hypercholesterolemia raised the hope that millions of Americans could avoid or postpone the development of heart disease. Because the interventions were potentially effective but were also costly, the cost-effectiveness of alternative approaches to detecting and treating hypercholesterolemia had become a critical issue for health policy.

The study was part of a three-grant initiative, Cost-Effective Strategies of Cholesterol-Lowering, which was recommended by the Arteriosclerosis, Hypertension, and Lipid Metabolism Advisory Committee in January, 1988 and given concept clearance at the September, 1988 National Heart, Lung, and Blood Advisory Council. The Request for Applications was released in March, 1990 and awards made in April, 1991.

DESIGN NARRATIVE:

Assessments were made of: effects of treatment on health outcomes (symptomatic coronary heart disease, death from coronary heart disease, and mortality from all causes); costs and effectiveness of specific dietary and pharmacological interventions; effects of delays in instituting treatment; effects of changing the interval between blood cholesterol tests on the probability and duration of treatment delay; cost and health consequences of modifying screening and treatment recommendations for other risk factors, age, and gender; population implications of screening and treatment strategies. Data from the Framingham Heart Study were used to estimate the time pattern of cholesterol levels, which was fundamental to the evaluation of changing the interval between cholesterol tests. Framingham data were also used to estimate the relation of event rates to blood cholesterol levels. Several components of the analysis were validated by testing model predictions against data from the Multiple Risk Factor Intervention Trial. The cost estimates were based on several additional sources. Individual-level cost-effectiveness estimates for several different interventions were presented along with population-level projections of the consequences of alternative strategies. The significance of altering assumptions about uncertain values, such as the long-term risks and benefits of specific medications, was tested in sensitivity analyses.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-04; Study Completion 1993-01

REFERENCES:
- [Background] Browner WS, Baron RB, Solkowitz S, Adler LJ, Gullion DS. Physician management of hypercholesterolemia. A randomized trial of continuing medical education. West J Med. 1994 Dec;161(6):572-8. PMID 7856157
- [Background] Hulley SB, Newman TB, Grady D, Garber AM, Baron RB, Browner WS. Should we be measuring blood cholesterol levels in young adults? JAMA. 1993 Mar 17;269(11):1416-9. PMID 8441219
- [Background] Garber AM, Browner WS, Hulley SB. Cholesterol screening in asymptomatic adults, revisited. Part 2. Ann Intern Med. 1996 Mar 1;124(5):518-31. doi: 10.7326/0003-4819-124-5-199603010-00013. PMID 8602715